CLINICAL TRIAL: NCT05824650
Title: Investigation of Activities of Daily Living, Cognition and Muscle Strength in Individuals With Frailty and Non-Fragile Congenital Heart Disease
Brief Title: Frailty and Non-Fragile Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Topcuoglu, Research Assistant, Hacettepe University
Other Study IDs: GO 23/20
Record Dates: First submitted 2023-03-29; First posted 2023-04-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Congenital Heart Disease; Frailty
Keywords: Congenital Heart Disease; Frailty
MeSH Terms: conditions — Heart Defects, Congenital; Frailty | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail Congenital Heart Disease Group: Frailty Fried et al. will be evaluated according to the five-parameter criteria set in the Cardiovascular Health Study by Having 3 or more parameters positive is defined as fragility. Individuals who meet this criterion will be included in this group.
  Interventions: Other: Observational
- Non-frail Congenital Heart Disease Group: Frailty Fried et al. will be evaluated according to the five-parameter criteria set in the Cardiovascular Health Study by Having 3 or more parameters positive is defined as fragility. Individuals who do not meet this criterion will be included in this group.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Individuals will be evaluated observationally in a 45-minute period in one day.

SUMMARY:
Congenital heart disease (CHD) is defined as congenital functional or anatomical abnormalities of the heart and intrathoracic great vessels. This study, which is planned to be carried out, will enable people with CHD to present a holistic perspective when planning rehabilitation programs and to create a common language for all health professionals.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is defined as congenital functional or anatomical abnormalities of the heart and intrathoracic great vessels. These abnormalities cover a wide range from minimal defects to serious cardiovascular problems. The prevalence of CHD has been reported as one case per 100 live births, with increases in recent years. As a result of surgical and medical advances in recent years, childhood lethal abnormalities in previous years can be significantly alleviated and repaired. As a result of these developments, 90% of patients born with CHD are expected to survive until adulthood, and today the number of adult CHD has exceeded the number of pediatric CHD. The aging CHD population is at risk of cardiovascular disease in addition to chronic problems resulting from congenital abnormalities. Frailty was defined by the Cardiovascular Health Study Collaborative Research Group as a complex clinical syndrome resulting from cumulative declines in more than one physiological system, leading to reduced resistance to risk factors. Loss of strength, decreased physical activity, involuntary weight loss, decreased mobility, and fatigue are sub-parameters of frailty. Frailty causes common pathophysiological mechanisms with risk factors that play a role in the development of cardiovascular disease. Frailty is associated with a higher incidence of cardiovascular disease and risks of all-cause mortality, leading to a reduction in life expectancy. Cardiorespiratory fitness and functional strength are shown to be the strongest predictors of frailty level and the potential for frailty to decrease over time. It has been reported that frailty worsens cognition and activities of daily living in cardiovascular diseases. There is no study in the literature that comprehensively evaluates vulnerability in individuals with CHD. The aim of this study; To assess frailty in individuals with CHD, to compare functional capacity, muscle strength, activities of daily living, and cognition in individuals with and without CHD. This study, which is planned to be carried out, will enable people with CHD to present a holistic perspective when planning rehabilitation programs and to create a common language for all health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital heart disease
* To be between the ages of 15-45
* To have been informed about the study and given written consent to participate in the study.

Exclusion Criteria:

* Having a neurological, orthopedic or any systemic disease,
* Presence of infection and malignancy,
* Cognitive, psychological and mental status are not suitable for evaluations,
* To undergo another surgery other than cardiac surgery.

Ages: 15 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: Congenital heart disease (CHD) is defined as congenital functional or anatomical abnormalities of the heart and intrathoracic great vessels. These abnormalities range from minimal defects to serious cardiovascular problems.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Frailty - Involuntary Weight Loss | 1 year
  Involuntary weight loss of more than 4.54 kg
Frailty - Loss of Strength | 1 year
  Grip strength will be evaluated using a grip dynamometer.
Frailty - International Physical Activity Questionnaire-Short Form | 1 week
  Physical activity assessment will be evaluated with the International Physical Activity Questionnaire-Short Form. The higher the score, the higher the physical activity; A low score indicates physical activity.
Frailty - Decreased mobility | 1 year
  It will be done with a walking test at a distance of 4 meters.
Frailty - Center for Epidemiologic Studies Depression Scale (CES-D). | 1 year
  Exhaustion was assessed by the Center for Epidemiologic Studies Depression Scale (CES-D). High scores indicate increased exhaustion; low scores indicate decreased exhaustion.
Functional capacity | 1 year
  Individuals will be asked to walk for 6 minutes at a distance of 30 meters
Peripheral Muscle Strength | 1 year
  Knee extensor and shoulder abductor muscle strength will be evaluated with digital dynamometer.
Daily Living Activities Evaluation | 1 year
  The Glittre Activities of Daily Living Test will be used to evaluate activities and functional status in daily life. Individuals start the test in a sitting position with backpacks weighing 5 kg for men and 2.5 kg for women. At a distance of 10 m between the chair and the shelf, when there is a 2-step ladder in the middle, patients must walk as quickly as possible and go up and down the steps, and take the one-kilogram bottles on the shelf first to the middle, then down, back to the middle, and finally up, and return, pass the step and sit on the chair. are asked to sit down and get up again, thus completing a round. Test completion time is recorded in minutes after completing five rounds
Montreal Cognitive Assessment Test | 1 year
  Cognition will be assessed by the Montreal Cognitive Assessment (MoCA) test. MoCA assesses functions such as short-term memory, visuospatial skills, executive functions, abstract thinking, verbal fluency, attention, concentration, and language. The highest total score that can be obtained from the test is 30. The normal limits of the test are 21 points and above. High scores increased cognitive function; low scores indicate decreased cognitive function.

SECONDARY OUTCOMES:
Body Composition | 1 year
  The lean body mass percentage of the individual will be determined by Bioelectrical Impedance Analysis. The measurement will be made by the individual standing on the device with bare feet and waiting. If the lean body mass percentage values are in the normal range, the body composition is normal; lean body mass percentage low values indicate deterioration of body composition.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No